CLINICAL TRIAL: NCT05455749
Title: A Prospective Pilot Study to Observe the Effects of Cat Exposure in an Allergen Exposure Chamber (AEC) in Cat Allergic Patients Taking a Food for Special Medical Purposes (holoBLG) for 3 Months
Brief Title: Effect of holoBLG on Cat Allergic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Allergy Therapeutics (Industry)
Collaborators: Ecarf Institute GmbH (Other); Bencard Allergie GmbH (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 039-P-21
Record Dates: First submitted 2022-07-08; First posted 2022-07-13 (Actual); Last update posted 2023-12-18 (Actual); Status verified 2022-07

CONDITIONS: Allergy to Cats; Allergic Rhinoconjunctivitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- holoBLG (Experimental)
  Interventions: Dietary Supplement: holoBLG

INTERVENTIONS:
Dietary Supplement: holoBLG — holo-BLG (beta-lactoglobulin) - a major component of the protein fraction of raw milk, loaded with ligands (vitamin A, zinc and polyphenol-iron complexes)

SUMMARY:
The aim of the study is to investigate the antigen-unspecific effect of a 3 months supplementation with a food for special medical purposes (FSMP) in form of a lozenge containing beta-lactoglobulin (BLG), iron, retinoic acid, zinc and polyphenols (holo-BLG) in patients with allergic rhinoconjunctivitis caused by cat (hair/dander) and the associated symptoms (symptom type and severity) during exposure to cat allergen in an Allergen Exposure Chamber (AEC).

ELIGIBILITY:
Inclusion Criteria:

* At least 1 year of clinically relevant cat allergy
* positive SPT (wheal >3mm)
* Positive NPT
* Increase in TSS >3 during the 1st exposure in the AEC
* Verbal and written consent

Exclusion Criteria:

* subjects <18 years
* subjects taking immunosuppressive drugs such as systemic corticosteroids, cyclosporine, etc.
* subjects who have received or are currently receiving sublingual or subcutaneous immunotherapy (SLIT/SCIT) for cat allergy in the last 2 years prior to V0
* clinically relevant overreactions to the ingredients of holoBLG, in particular subjects with a milk protein allergy or pronounced lactose intolerance
* subjects with severe asthma and/or a history of uncontrolled asthmatic attacks in the last three months before the selection process (GINA 4 and 5).
* subjects with an FEV1 <70% (predicted value) prior to exposure in the AEC
* Lack of verbal and written informed consent
* subjects who are not proficient in the German language
* History of serious chronic medical illness and/or any condition for which the local investigator believes that participation in the study could pose a risk to the individual
* Pregnancy and lactation
* Contraindications and/or history of adrenaline intolerance and/or emergency medications
* Concurrent use of anti-allergic medications and/or inadequate washout period of these anti-allergic medications prior to the selection process and exposure in the exposure chamber
* TSS ≥ 6 at t0 of first exposure in the AEC
* Subjects who have a history of ingestion of holoBLG

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2021-10-04 (Actual); Primary Completion 2022-03-15 (Actual); Study Completion 2022-03-16 (Actual)

PRIMARY OUTCOMES:
TSS | After 120 minutes of allergen challenge
  Total Symptom Score in response to cat exposure in an AEC at baseline versus final AEC exposure. The TSS is the sum of 4 nose symptoms (runny nose, sneezing, itchy nose, and blocked nose), 4 eye symptoms (itchy eyes, watery eyes, gritty feeling, eye reddening), 4 bronchial symptoms (wheezing, cough, breathlessness, rhonchus), and 2 other symptoms (itchy palate, and itchy skin) on a scale of 0 to 3 (no symptoms, mild symptoms, moderate symptoms, and severe symptoms), leading to a maximum TSS of 42.

SECONDARY OUTCOMES:
TNSS | Up to 120 minutes following allergen challenge
  The Total Nasal Symptom Score (TNSS) is the sum of 4 nose symptoms (runny nose, sneezing, itchy nose, and blocked nose) on a scale of 0 to 3 (no symptoms, mild symptoms, moderate symptoms, and severe symptoms), leading to a maximum TNSS of 12.
TESS | Up to 120 minutes following allergen challenge
  The Total Eye Symptom Score (TESS) is the sum of 4 eye symptoms (itchy eyes, watery eyes, gritty feeling, eye reddening) on a scale of 0 to 3 (no symptoms, mild symptoms, moderate symptoms, and severe symptoms), leading to a maximum TESS of 12.
TBSS | Up to 120 minutes following allergen challenge
  The Total Bronchial Symptom Score (TBSS) is the sum of 4 bronchial symptoms (wheezing, cough, breathlessness, rhonchus) on a scale of 0 to 3 (no symptoms, mild symptoms, moderate symptoms, and severe symptoms), leading to a maximum TBSS of 12.
VAS | Recorded at time zero (0) and every 30 minutes during exposure until 120 minutes
  Visual Analogue Scale: Before, every 30 minutes during and after each exposure patients grade the question on their well-being by putting a vertical line on a 10 cm line representing severity from 0 cm "very good" to 10 cm "very bad".
PNIF | Recorded at time zero (0) and every 30 minutes during allergen exposure up to 120 minutes
  PNIF (peak nasal inspiration flow) liter/minute.
PEF | Recorded at time zero (0) and every 30 minutes during allergen exposure up to 120 minutes
  PEF (peak expiratory flow) liter/minute
FEV1 | Recorded at time zero (0) and 120 minutes
  Forced expiratory volume in 1 second, before and after the exposure
FEV1/FVC | Recorded at time zero (0) and 120 minutes
  Forced expiratory volume in 1 second/forced vital capacity ratio, before and after the exposure.
Adverse events with regards to the allergen exposure | up to 24 hours after AEC exposure
  Number of events and number of patients recording late-phase reactions and/or adverse events with regards to the allergen exposure
NPT | up to 3 months following first AEC
  Changes in Nasal Provocation Test before and after intervention period
TOSS | Up to 120 minutes following allergen challenge
  The Total Other Symptom Score (TBSS) is the sum of 2 additional symptoms (itchy palate, itchy skin) on a scale of 0 to 3 (no symptoms, mild symptoms, moderate symptoms, and severe symptoms), leading to a maximum TOSS of 6.

CONTACTS AND LOCATIONS:
Overall Officials: Karl-Christian Bergmann, Prof. Dr. med., Principal Investigator — Institute of Allergology, Charité - Universitätsmedizin Berlin, corporate member of Freie Universität Berlin and Humboldt-Universität zu Berlin, Berlin, Germany
Locations (1):
- ECARF Institute GmbH, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bergmann KC, Raab J, Graessel A, Zwingers T, Becker S, Kugler S, Zuberbier T, Roth-Walter F, Kramer MF, Jensen-Jarolim E. The holo beta-lactoglobulin lozenge reduces symptoms in cat allergy-Evaluation in an allergen exposure chamber and by titrated nasal allergen challenge. Clin Transl Allergy. 2023 Jul;13(7):e12274. doi: 10.1002/clt2.12274. PMID 37488734